CLINICAL TRIAL: NCT00468143
Title: A Within-Subject Cross-Over Comparison Between Immediate Release and Extended Release Adderall
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IR v XR
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Results first posted 2016-06-02 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Adderall; SLI381

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adderall Extended Release First (Experimental): This group was treated with Adderall extended release, either during phase 2 of the trial, or during phase 3 (this subset received Adderall immediate release during phase 2 and then underwent a washout period). This was a counterbalanced crossover study, with a washout period in between treatment periods. Participants were randomized in a 1:1 ratio to one of two schedules Adderall IR followed by Adderall XR, or Adderall XR followed by Adderall IR.
  Interventions: Drug: Adderall ® Immediate Release; Drug: Adderall XR ®
- Adderall Immediate Release First (Experimental): This group was treated with Adderall immediate release, either during phase 2 of the trial, or during phase 3 (this subset received Adderall extended release during phase 2 and then underwent a washout period). This was a counterbalanced crossover study, with a washout period in between treatment periods. Participants were randomized in a 1:1 ratio to one of two schedules Adderall IR followed by Adderall XR, or Adderall XR followed by Adderall IR.
  Interventions: Drug: Adderall ® Immediate Release; Drug: Adderall XR ®

INTERVENTIONS:
Drug: Adderall ® Immediate Release — Adderall Immediate release (IR) was provided as treatment for three weeks (at 15, 30 or 45 mg TID). The medication was optimized for titration.
Drug: Adderall XR ® — Adderall Extended Release (XR) was provided as treatment for three weeks at (15, 30, or 45 mg QD). The medication was optimized for titration.
  Other Names: extended release adderall

SUMMARY:
The purpose of this pilot study is to compare Adderall ® and Adderall XR ® in terms of their effectiveness and side effects for the treatment of ADHD in adults.

DETAILED DESCRIPTION:
This will be a randomized, cross-over study in which adults with ADHD will receive three weeks of treatment with Adderall (IR) (15, 30, or 45 mg TID) and three weeks of treatment of Adderall XR (XR) (15, 30, or 45 mg QD) for evaluation of dosing adherence and treatment efficacy. The order of the two conditions (TID-QD or QD-TID) will be counterbalanced across subjects, with a washout period in between treatment periods. Participants will be required to come to the site for 9 visits over approximately an 8-week period.

The study will consist of the following four phases:

* Phase 1

  * Screening Visit (Visit 1)
  * Treatment "A" Baseline Visit (Visit 2)
* Phase 2

  o Treatment Period "A" - participants will take either Adderall or Adderall XR for 3 weeks (Visits 3-5)
* Phase 3

  * 7-Day Washout Period - participants will be off Treatment "A" medication
  * Treatment "B" Baseline visit (Visit 6)
* Phase 4 o Treatment Period "B" - participants will take either Adderall or Adderall XR for 3 weeks (Visits 7-9)

Eligible participants will be randomized in a 1:1 ratio to one of two schedules of treatment, Adderall IR followed by Adderall XR, or Adderall XR followed by Adderall IR. Within both schedules, each treatment will consist of a 3-week dose optimization titration evaluation period with a washout week prior to switching to the second respective treatment. The maximum total daily dose will be 45mg, with 15mg TID for IR or 45mg QD for XR. Throughout the medication treatment periods, participants will visit the clinic weekly for evaluations of efficacy, tolerance, and adherence. Medical evaluations will also be conducted at each treatment visit, including assessment of weight, blood pressure, and pulse. Efficacy and adherence data will collected by separate research staff, so that the rater evaluating efficacy will be blinded to the adherence results. The clinician evaluating efficacy will also be blinded to the participants' treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of consent, are between the ages of 18-55, inclusive.
2. Meet DSM-IV criteria for ADHD as assessed by the Adult ADHD Clinician Diagnostic Scale (ACDS) v1.2.
3. Female participants of childbearing potential must test negative for pregnancy at the time of enrollment based on a urine pregnancy test and agree to use a reliable method of birth control during the study. Females of childbearing potential are defined as women not surgically sterilized and are between menarche and 2 years post-menopause.
4. Must have a satisfactory medical assessment with no clinically significant abnormalities as determined by medical history, physical exam, ECG, and clinical laboratory testing.
5. Must be able to swallow capsules.
6. Must be able to begin the daily dose of study medication in the morning.
7. Must be off previous amphetamine or methylphenidate treatment for 1 week prior to baseline (visit 2). Must be off past non-stimulant ADHD medication (i.e., atomoxetine) for 3 weeks prior to baseline (visit 2).
8. In the opinion of the investigator, the subject must understand and be able, willing and likely to fully comply with the study procedures and restrictions.
9. Must have given signed and dated informed consent in accordance with Good Clinical Practice (GCP) Guidelines.

Exclusion Criteria:

1. Lifetime or present history of bipolar disorder, schizophrenia or schizoaffective disorder.
2. Uncontrolled comorbid major depressive disorder, anxiety disorder or dysthymia. Participants with controlled depressive or anxiety disorders may participate if their medications have been stabilized for a minimum of four weeks and, in the opinion of the Principal Investigator, will not interfere with adherence, safety, or efficacy assessments.
3. Anyone who meets current DSM-IV-TR criteria for alcohol or any non-alcohol substance abuse or dependence disorder (excluding nicotine).
4. Have organic brain disease (such as dementia) or traumatic brain injury residua. Have a history of seizure disorder (other than febrile seizures) or participants who have taken (or are currently taking) anticonvulsants for seizure control.
5. Females who are currently pregnant or breast feeding, and women of child-bearing potential who are not currently using an adequate form of birth control.
6. Participants with clinically significant ECG or laboratory abnormalities at screening that are deemed exclusionary in the opinion of the Principal Investigator.
7. Participants who work the night shift or another schedule that would preclude beginning the daily dose of study medication in the morning.
8. Participants with a positive urine drug result at Screening.
9. Participants with any concurrent chronic or acute illness or unstable medical condition that could, in the opinion of the study physician, confound the results of safety assessments, increase risk to the subject or lead to difficulty complying with the protocol. Subjects who have a history of mental retardation or severe learning disability will be excluded.
10. Participants with a history of structural cardiac abnormalities as well as any other condition that may affect cardiac performance.
11. Participants with documented history of allergy, intolerance, or non-responsivity to methylphenidate or amphetamines. This includes a history of two or more failed stimulant treatment trials, as deemed by the Principal Investigator.
12. Participants who in the investigator's opinion meet any of the exclusionary criteria specified on the FDA label of either Adderall or Adderall XR.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2007-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lenard Adler, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- VANYHHS, New York, New York, United States

REFERENCES:
- [Derived] Adler LA, Lynch LR, Shaw DM, Wallace SP, Ciranni MA, Briggie AM, Kulaga A, O'Donnell KE, Faraone SV. Medication adherence and symptom reduction in adults treated with mixed amphetamine salts in a randomized crossover study. Postgrad Med. 2011 Sep;123(5):71-9. doi: 10.3810/pgm.2011.09.2461. PMID 21904088

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men or women, aged 18 to 55 years, who met the DSM-IV criteria for ADHD, as assessed by the Adult ADHD Clinician Diagnostic Scale (ACDS) version 1.2, were eligible to participate. Participants were recruited from local advertising or from the pool of participants at the MHADRP at NYU School of Medicine and VA NY Harbor Healthcare System.
Pre-assignment Details: Individuals who were currently receiving amphetamine or methylphenidate treatment underwent a 7-day washout period before the baseline visit; those receiving atomoxetine or other medications for ADHD were required to undergo a 28-day washout period before the baseline visit. While 62 subjects started the study, only 49 finished the full study.
Groups:
- Extended Release First: This group received the extended release medication during the first three weeks of treatment and then received the immediate release medication during the last 3 weeks of treatment.
- Immediate Release First: This group received the immediate release medication during the first three weeks of treatment and then received the extended release medication during the last 3 weeks of treatment.
Period: First Intervention (3 Weeks)
Arm/Group | Extended Release First | Immediate Release First
Started | 31 | 31
Completed | 28 | 27
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 4
Period: Second Intervention (3 Weeks)
Arm/Group | Extended Release First | Immediate Release First
Started | 28 | 27
Completed | 25 | 24
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- All Participants: This was a randomized, crossover study in which participants received 3 weeks of treatment with MAS IR (15, 30, or 45 mg TID) and 3 weeks of treatment with MAS XR (15, 30, or 45 mg qAM). The order of the treatments (TID-qAM or qAM-TID) was counterbalanced across participants, with a washout period of ≥ 7 days between epochs.
Arm/Group | All Participants
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 34
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 46
  African American | 7
  Hispanic | 5
  Asian | 4

OUTCOME MEASURES:

1. Primary Outcome: Medication Event Monitoring System (MEMS®) Dosage Adherence
Description: Dosage adherence (MEMSd) is the number of bottle openings divided by number of doses prescribed. Adherence was measured as ≥ 75% of the doses. The number below is the total percentage of subjects who were adherent.
Time Frame: The MEMS information was noted at clinic visit 3, 4, 5, 7, 8, and 9 (over 8 weeks)
Population: These is the total of participants who completed the study.
Measure: Number; unit: percentage of participants adherent
Groups:
- Adderall IR (Methamphetamine Salts): All participants were initiated at a total daily dose of 15 mg/day (5 mg TID for Adderall IR (Methamphetamine Salts)). At visits 3 and 4, the total daily dose of MAS was increased by 15 mg/day until an optimal dose or the maximum total daily dose of 45 mg/day was reached. An optimal dose was determined by clinical efficacy (a ≥ 30% reduction in the baseline total ADHD Rating Scale [ADHD-RS] scores) and tolerability.
- Adderall XR (Methamphetamine Salts): All participants were initiated at a total daily dose of 15 mg/day (15 mg qAM for Adderall XR (Methamphetamine Salts)). At visits 3 and 4, the total daily dose of MAS was increased by 15 mg/day until an optimal dose or the maximum total daily dose of 45 mg/day was reached. An optimal dose was determined by clinical efficacy (a ≥ 30% reduction in the baseline total ADHD Rating Scale [ADHD-RS] scores) and tolerability.
Arm/Group | Adderall IR (Methamphetamine Salts) | Adderall XR (Methamphetamine Salts)
Number analyzed (Participants) | 49 | 49
percentage of participants adherent | 42.7 | 66.2

2. Primary Outcome: Medication Event Monitoring System (MEMS®) Regimen Adherence
Description: Regimen adherence (MEMSr) is a percentage of the number of days in which the complete dose regimen was taken as prescribed. Adherence was measured as complete dose regimen taken on ≥ 90% of days. The number below is the total percentage of subjects who were adherent.
Time Frame: The MEMS information was noted at clinic visit 3, 4, 5, 7, 8, and 9 (over 8 weeks)
Measure: Number; unit: percentage of participants adherent
Arm/Group | Adderall IR (Methamphetamine Salts) | Adderall XR (Methamphetamine Salts)
Number analyzed (Participants) | 49 | 49
percentage of participants adherent | 2.5 | 34.4

3. Primary Outcome: Medication Event Monitoring System (MEMS®) Time Adherence
Description: Time adherence (MEMSt) is the percentage of doses taken as prescribed within a specified time period. Adherence was measured as ≥ 80% of doses taken at the correct time. The number below is the percentage of subjects who were adherent.
Time Frame: The MEMS information was noted at clinic visit 3, 4, 5, 7, 8, and 9 (over 8 weeks)
Measure: Number; unit: percentage of participants adherent
Arm/Group | Adderall IR (Methamphetamine Salts) | Adderall XR (Methamphetamine Salts)
Number analyzed (Participants) | 49 | 49
percentage of participants adherent | 4.5 | 43.7

4. Secondary Outcome: Pill Count
Description: Study staff counted unused medication at each weekly visit to yield a percentage of prescribed pills that were consumed. For each group, the number given will be the total number of consumed pills divided by total number of pill prescribed.
Time Frame: At clinic visit 3, 4, 5, 7, 8, and 9 (over 8 weeks)
Measure: Number; unit: percentage of pills consumed
Arm/Group | Adderall IR (Methamphetamine Salts) | Adderall XR (Methamphetamine Salts)
Number analyzed (Participants) | 49 | 49
percentage of pills consumed | 90.4 | 96.9

5. Secondary Outcome: Self Report
Description: Self-reported adherence was ascertained via retrospective self-report of daily regimen adherence. Participants were considered adherent for Adderall IR (Methamphetamine salts) if they took the first does in the morning within 30 minutes of waking, and then each subsequent dose in 5-hour intervals (within 30 minutes). For Adderall XR (Methamphetamine salts), participants were considered adherent if they took the single daily dose in the morning within 30 minutes of waking. The number given below represents the total number of self-reported adherent participants divided by the total number of participants per group, times 100 (to obtain percentage).
Time Frame: At clinic visit 3, 4, 5, 7, 8, and 9 (over 8 weeks)
Measure: Number; unit: percentage of participants adherent
Arm/Group | Adderall IR (Methamphetamine Salts) | Adderall XR (Methamphetamine Salts)
Number analyzed (Participants) | 49 | 49
percentage of participants adherent | 92.6 | 98.8

ADVERSE EVENTS:
Groups:
- Extended Release; Immediate Release: This was a randomized, crossover study in which participants received 3 weeks of treatment with MAS IR (15, 30, or 45 mg TID) and 3 weeks of treatment with MAS XR (15, 30, or 45 mg qAM). The order of the treatments (TID-qAM or qAM-TID) was counterbalanced across participants, with a washout period of ≥ 7 days between epochs.
Arm/Group | Extended Release | Immediate Release
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 53/62 | 53/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Release (N=62) | Immediate Release (N=62)
Headache (Vascular disorders) | 4 (6) | 11 (11)
Insomnia (General disorders) | 14 (15) | 19 (20)
Loss of Appetite/Anorexia (General disorders) | 23 (26) | 5 (7)
Anxiety (Psychiatric disorders) | 7 (8) | 4 (6)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Feeling Speedy or Wired or Jittery (Psychiatric disorders) | 6 (6) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dry Mouth (General disorders) | 14 (15) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No